CLINICAL TRIAL: NCT01223599
Title: Rhomboid Flap Versus Primary Closure
Brief Title: Rhomboid Flap Versus Primary Closure After Excision of Sacrococcygeal Pilonidal Sinus. (A Prospective Randomized Study)
Acronym: non
Status: Withdrawn | Type: Observational
Sponsor: Mansoura University (Other)
Other Study IDs: non
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Evaluate and Compare Between Excision and Primary Closure Procedure and Rhomboid Flap Technique for the Treatment of Pilonidal Sinus; Duration of Operation,
Keywords: pilonidal disease; natal cleft; limberg flap

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To evaluate and compare between excision with primary closure of wound and excision with Rhomboid flap reconstruction in the treatment of pilonidal sinus as regard duration of operation, healing time, hospital stay, complications and recurrence rate.

ELIGIBILITY:
Inclusion Criteria:

* chronic pilonidal sinus

Exclusion Criteria:

* pilonidal abcess

Ages: 15 Years to 43 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: both sex different age april 2008-march 2010
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2008-04; Study Completion 2010-03